CLINICAL TRIAL: NCT04806321
Title: Project SOLVE: A School-based Trial of a Universal Single-session Digital Problem-solving Intervention for Adolescent Mental Health
Brief Title: Project SOLVE: Trial of a Brief Digital Problem-solving Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Responsible Party: Principal Investigator, Olivia Fitzpatrick, Principal Investigator; Doctoral Student, Harvard University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB20-1791
Record Dates: First submitted 2021-03-08; First posted 2021-03-19 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Anxiety; Depression; Stress
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Participants (anticipated N = 1,000), ages 10-14 years old, will be randomized to complete one of two 30-minute, digital programs: (1) Project SOLVE: a program designed to teach adolescents how to solve, rather than be overwhelmed by, everyday problems; or (2) Project SUCCESS: a control program designed to teach adolescents helpful study skills.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Project SOLVE (Experimental): This program is self-guided, digital, and approximately 30 minutes in length. Content is designed to help adolescents solve, rather than be overwhelmed by, everyday problems. The program includes: (1) An introduction to problem solving; (2) Testimonials from "valued others" (older adolescents; celebrities) describing their use of problem solving skills; (3) Evidence from studies that our brains are capable of problem solving and that problem solving can be helpful; and (4) Activities designed to enable adolescents to practice sequential problem solving using a few steps (SOLVE Steps).
  Interventions: Other: Project SOLVE
- Project SUCCESS (Active Comparator): This program is self-guided, digital, and approximately 30 minutes in length. Content is designed to help adolescents improve their study skills. This program includes: (1) An introduction to study skills; (2) Testimonials from "valued others" describing their use of study skills; (3) Description of helpful and commonly used study skills (e.g., note-taking); and (4) Activities designed to encourage adolescents to practice these skills in their daily lives.
  Interventions: Other: Project SUCCESS

INTERVENTIONS:
Other: Project SOLVE — This 30-minute, self-guided, digital program is designed to help adolescents solve, rather than be overwhelmed by, everyday problems.
  Arms: Project SOLVE
Other: Project SUCCESS — This 30-minute, self-guided, digital program is designed to help adolescents develop study skills.
  Arms: Project SUCCESS

SUMMARY:
The goal of this trial is to examine the effectiveness of a universal, self-guided, digital single-session intervention focusing on problem-solving skills in improving adolescent mental health and well-being, relative to an active control intervention focusing on study skills, within the context of school settings during the coronavirus disease pandemic.

DETAILED DESCRIPTION:
More than 20% of adolescents will experience at least one mental health disorder or problem before adulthood that warrants treatment, yet 80% of these adolescents will never receive care. This need-to-access gap appears to be heightened during the current coronavirus disease pandemic and its resulting disruptions to healthcare and education systems. Both within and beyond the context of the pandemic, preventive mental health interventions are positioned to help adolescents build and strengthen coping strategies that can preclude the emergence of mental health difficulties that require more resource-intensive levels of clinical care. Preventive mental health interventions delivered via digital platforms and within school-based settings might be especially scalable.

The current school-based trial is designed to test one such strategy that harnesses technology to boost the scalability of adolescent mental health interventions: a brief (one 30 minute session) digital program designed to empower adolescents (10-14 years old) to solve, rather than be overwhelmed by, everyday problems (Project SOLVE). Single-session interventions designed to help adolescents cultivate adaptive mindsets have reduced anxiety and depression among adolescents with and without elevated symptoms of these disorders. Building on this strong foundation, Project SOLVE targets these mental health challenges with problem solving skills-one of the most versatile, commonly used, and potent therapeutic techniques for adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent is in grades 6-8 (inclusive) at partnering schools
* Adolescent is between the ages of 10-14 years (inclusive) at the time of study enrollment
* Adolescent and at least one guardian consent to adolescent participation in study
* Adolescent reads English well enough to effectively complete the digital programs
* Adolescent has access to a digital device

Exclusion Criteria:

* Adolescent is non-English speaking, as the programs are only available in English
* Adolescent does not have access to a digital device
* Adolescent has an intellectual disability that precludes comprehension of the program content

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 522 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Change in Behavior and Feelings Survey (Internalizing Subscale) From Baseline to 3-month Follow-Up | Baseline to 3-month follow-up
  Trajectories of self-reported symptoms of anxiety and depression from the 6-item (each item rated on a 0-4 scale, with higher ratings indicating more symptoms) Internalizing subscale of the Behavior and Feelings Survey. Total scores range from 0 to 24, with higher scores indicating more symptoms.
Change in Behavior and Feelings Survey (Internalizing Subscale) From Baseline to 12-month Follow-Up | Baseline to 12-month follow-up
  Trajectories of self-reported symptoms of anxiety and depression from the 6-item (each item rated on a 0-4 scale, with higher ratings indicating more symptoms) Internalizing subscale of the Behavior and Feelings Survey. Total scores range from 0 to 24, with higher scores indicating more symptoms.
Change in State Hope Scale Pathways Subscale From Immediately Pre-Intervention to Immediately Post-Intervention | Immediately pre-intervention to immediately post-intervention
  Change in self-reported hopefulness, as measured via the 3-item "pathways" (planning of ways to meet goals) subscale of the State Hope Scale. Each item is rated on a 1-8 scale and total scores range from 1 to 24, with higher scores indicating higher levels of hopefulness.
Change in Beck Hopelessness Scale From Immediately Pre-Intervention to Immediately Post-Intervention | Immediately pre-intervention to immediately post-intervention
  The Beck Hopelessness Scale (BHS) asks adolescents to rate 4 statements based on their sense of hopelessness. Participants rate the 4 statements on a 4 point scale ranging from 0 (Absolutely Disagree) to 3 (Absolutely Agree). Total score ranges from 0 to 12, with higher scores indicating greater levels of hopelessness.

SECONDARY OUTCOMES:
Perceived Program Acceptability and Helpfulness | Immediately post-intervention
  Post-intervention feedback on the program's perceived acceptability and helpfulness as measured via a 7-item scale, with each item rated on a 1-5 scale, with higher scores indicating greater acceptability and helpfulness.
Change in Behavior and Feelings Survey (Externalizing Subscale) From Baseline to 3-month Follow-Up | Baseline to 3-month follow-up
  Trajectories of self-reported misbehavior from the 6-item (each item rated on a 0-4 scale, with higher ratings indicating more symptoms) Externalizing subscale of the Behavior and Feelings Survey. Total scores range from 0 to 24, with higher scores indicating more symptoms.
Change in Behavior and Feelings Survey (Externalizing Subscale) From Baseline to 12-month Follow-Up | Baseline to 12-month follow-up
  Trajectories of self-reported misbehavior from the 6-item (each item rated on a 0-4 scale, with higher ratings indicating more symptoms) Externalizing subscale of the Behavior and Feelings Survey. Total scores range from 0 to 24, with higher scores indicating more symptoms.
Change in State Hope Scale From Baseline to 3-Month Follow-Up | Baseline to 3-month follow-up
  Change in self-reported total hopefulness from the 6-item (each item rated on a 1-8 scale, with higher scores indicating greater hopefulness) State Hope Scale, as well as self-reported scores on the 3-item "agency" (goal-directed determination) and 3-item "pathways" (planning of ways to meet goals) subscales of this measure.
Change in State Hope Scale From Baseline to 12-Month Follow-Up | Baseline to 12-month follow-up
  Change in self-reported total hopefulness from the 6-item (each item rated on a 1-8 scale, with higher scores indicating greater hopefulness) State Hope Scale, as well as self-reported scores on the 3-item "agency" (goal-directed determination) and 3-item "pathways" (planning of ways to meet goals) subscales of this measure.
Change in Beck Hopelessness Scale From Baseline to 3-Month Follow-Up | Baseline to 3-month follow-up
  The Beck Hopelessness Scale (BHS) asks adolescents to rate 4 statements based on their sense of hopelessness. Participants rate the 4 statements on a 4 point scale ranging from 0 (Absolutely Disagree) to 3 (Absolutely Agree). Total score ranges from 0 to 12, with higher scores indicating greater levels of hopelessness.
Change in Beck Hopelessness Scale From Baseline to 12-Month Follow-Up | Baseline to 12-month follow-up
  The Beck Hopelessness Scale (BHS) asks adolescents to rate 4 statements based on their sense of hopelessness. Participants rate the 4 statements on a 4 point scale ranging from 0 (Absolutely Disagree) to 3 (Absolutely Agree). Total score ranges from 0 to 12, with higher scores indicating greater levels of hopelessness.

CONTACTS AND LOCATIONS:
Locations (1):
- Harvard University, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Analytic code will be made available upon publication of trial results. Study protocol and SAP are available with this registration submission.

REFERENCES:
- [Derived] Steinberg JS, Fitzpatrick OM, Khurana S, Kim MY, Mair P, Schleider JL, Hatzenbuehler ML, Weisz JR. Is There a Place for Cognitive Restructuring in Brief, Self-Guided Interventions? Randomized Controlled Trial of a Single-Session, Digital Program for Adolescents. J Clin Child Adolesc Psychol. 2024 Aug 9:1-21. doi: 10.1080/15374416.2024.2384026. Online ahead of print. PMID 39120779

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-20): https://cdn.clinicaltrials.gov/large-docs/21/NCT04806321/Prot_SAP_000.pdf